CLINICAL TRIAL: NCT05507879
Title: Characterization of TRPC6 to Predict and Prevent Chemotherapy Related Cardiomyopathy and Heart Failure (Prospective Study)
Brief Title: TRPC6 Characterization to Predict and Prevent Chemotherapy Related Cardiomyopathy and Heart Failure With Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-001501; NCI-2022-05690 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); W81XWH-22-1-0289 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-08-08; First posted 2022-08-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Carcinoma; Cardiomyopathy; Congestive Heart Failure
MeSH Terms: conditions — Breast Neoplasms; Cardiomyopathies; Heart Failure | interventions — Specimen Handling; Electronic Health Records

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biospecimen collection): Patients undergo collection of blood samples at time of therapy initiation. Patients who develop cardiac toxicity may undergo additional collection of blood samples. Patients' medical records are also reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Medical Record

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Medical Record — Review of medical records
  Other Names: Computer Based Patient Record; EMR; EMR (electronic medical record)

SUMMARY:
This study examines TRPC6 in predicting and preventing chemotherapy related cardiac toxicity and heart failure in patients with breast cancer. Cardiac toxicity, changes in heart function is a well-recognized complication of certain cancer related therapies. Understanding these changes may allow early intervention against therapy-related cardiac toxicity and also identify novel therapeutic targets to protect patient long-term cardiac health. Studying samples of blood from patients with breast cancer in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA), identify biomarkers related to cardiac toxicity, and prevent the development of therapy-induced cardiac toxicity in patients receiving chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Characterize TRPC6 risk variants for doxorubicin-related cardiotoxicity in prospectively collected samples from breast cancer patients.

OUTLINE: This is an ancillary-correlative study.

Patients undergo collection of blood samples at time of enrollment. Patients who develop cardiac toxicity may undergo additional collection of blood samples. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Any breast cancer patient initiating doxorubicin/other anthracycline and patients receiving trastuzumab without doxorubicin/anthracycline in the neoadjuvant/adjuvant setting
* An understanding of the protocol and its requirements, risks, and discomforts
* The ability and willingness to sign an informed consent
* Diagnosed with therapy related cardiotoxicity defined as; cardiomyopathy, symptomatic heart failure, asymptomatic reduced systolic function, acute coronary syndrome, myocardial infarction, critical limb ischemia, cardiac arrhythmias or myocarditis possibly related to prior cancer treatment OR completed chemotherapy with no cardiotoxicity at least two years post treatment OR patients with cancer who will be initiating systemic therapy with potentially cardiotoxic medications. This will include doxorubicin chemotherapy, or trastuzumab.
* Healthy, non-pregnant, adult subjects who weigh at least 110 pounds

Exclusion Criteria:

* Inability on the part of the patient to understand the informed consent or be compliant with the protocol
* Anemia with hemoglobin less than 8
* Patients not willing to undergo a blood draw
* Patients with stage IV or distant metastatic breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer who have previously received chemotherapy, are currently being treated with chemotherapy, or are about to be treated with chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Significance ofTRPC6 coding sequencing | Up to study completion, up to four years to completion.
  Will compare the prevalence of rare missense variants in our cases against the null hypothesis to assess the significance of TRPC6 coding sequencing data in patients with dox-induced heart failure (HF). Will use an exploratory analysis to estimate the prevalence, 95% confidence intervals and p-values depending on the number of patients with rare variants in the data set and due to the rarity (i.e. high degree of conservation in the TRPC6 coding sequence).Other methods include biospecimen collection and the TRPC6 coding sequence. Data collected will be stored in a database and studied by the PI.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Norton, Ph.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials